CLINICAL TRIAL: NCT05569954
Title: A Phase 3, Randomized, Double-blind, Active Comparator-controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Adults 50 Years of Age or Older
Brief Title: Safety and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Adults 50 Years of Age or Older (V116-010, STRIDE-10)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V116-010; 2022-503144-40-00 (Registry Identifier: EU CT); U1111-1286-5378 (Registry Identifier: UTN); 2022-001785-35 (EudraCT Number)
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V116 (Experimental): Participants will receive a single intramuscular (IM) vaccination of 0.5 mL of V116 on Day 1.
  Interventions: Biological: V116
- PPSV23 (Active Comparator): Participants will receive a single IM vaccination of 0.5 mL of PPSV23 on Day 1.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Sterile 0.5 mL solution in prefilled syringe containing 4 μg of each pneumococcal polysaccharide (PnPs) antigen 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B.
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116
Biological: PPSV23 — Sterile 0.5 mL solution in prefilled syringe containing 25 μg of each PnPs antigen 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F.
  Other Names: PNEUMOVAX™23
  Arms: PPSV23

SUMMARY:
This is a phase 3, randomized, double-blind, active comparator-controlled study of the safety, tolerability, and immunogenicity of V116 in pneumococcal vaccine-naïve adults 50 years of age and older. The polyvalent (23-valent) pneumococcal vaccine, PPSV23, is the active comparator. In addition to studying safety/tolerability, it is hypothesized that, at 30 days postvaccination, the immunogenicity of V116 is noninferior to PPSV23 for the 12 common serotypes in V116 and PPSV23, and that V116 is superior to PPSV23 for the 9 serotypes unique to V116. It is also hypothesized that V116 is superior to PPSV23 in the percentage of participants with ≥4-fold rise from baseline in unique V116 serotypes, as measured by serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs).

DETAILED DESCRIPTION:
Selected participants may be eligible for optional immunogenicity or PBMC substudies extension that will investigate the exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

* For females, is not pregnant or breastfeeding and is either not a woman of childbearing potential (WOCBP) or is a WOCBP and uses acceptable contraception/abstinence; and has medical, menstrual, and recent sexual activity history reviewed by the investigator to decrease the chance of inclusion of an early undetected pregnancy

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD) [positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site] or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1)
* Has a known hypersensitivity to any component of V116 or PPSV23, including diphtheria toxoid
* Has a known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating IM vaccination
* Had a recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring <72 hours before receipt of study vaccine
* Has a known malignancy that is progressing or has required active treatment <3 years before enrollment
* Received prior pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside the protocol
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention ≥14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received any nonlive vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any nonlive vaccine ≤30 days after receipt of study vaccine (inactivated influenza and SARS-CoV2 vaccines may be acceptable)
* Received any live virus vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of study vaccine
* Received a blood transfusion or blood products, including immunoglobulin ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product until the Day 30 postvaccination blood draw is complete

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1484 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2025-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (55):
- Fundacion Estudios Clinicos ( Site 0200), Rosario, Santa Fe Province, Argentina
- Australia (3):
  - Paratus Clinical Research Western Sydney ( Site 1500), Blacktown, New South Wales
  - Northern Beaches Clinical Research ( Site 1502), Brookvale, New South Wales
  - Paratus Clinical Research Brisbane ( Site 1501), Albion, Queensland
- Colombia (2):
  - IPS Centro Científico Asistencial S.A.S ( Site 0407), Barranquilla, Atlántico
  - Fundacion Valle del Lili- CIC ( Site 0415), Cali, Valle del Cauca Department
- Germany (5):
  - klinikum rechts der isar der technischen universität münchen ( Site 0904), München, Bavaria
  - InfektioResearch ( Site 0903), Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln ( Site 0900), Cologne, North Rhine-Westphalia
  - Medizentrum Essen Borbeck ( Site 0902), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf-Infektiologie ( Site 0901), Hamburg
- Israel (5):
  - Rambam Health Care Campus ( Site 1002), Haifa
  - Hadassah Medical Center-Clinical Reaserch Unit ( Site 1004), Jerusalem
  - Meir Medical Center-Infectious unit ( Site 1003), Kfar Saba
  - Sheba Medical Center ( Site 1000), Ramat Gan
  - Clalit Health Services - Sakhnin Community Clinic-Research Unit ( Site 1001), Sakhnin
- New Zealand (3):
  - P3 Research - Palmerston North ( Site 1602), Palmerston North, Manawatu-Wanganui
  - P3 Research - Lower Hutt ( Site 1601), Lower Hutt, Wellington Region
  - Optimal Clinical Trials ( Site 1600), Auckland
- South Korea (15):
  - Wonju Severance Christian Hospital ( Site 1808), Wŏnju, Kang-won-do
  - Chonnam National University Hospital-Infectious Diseases ( Site 1811), Gwangju, Kwangju-Kwangyokshi
  - Korea University Ansan Hospital ( Site 1801), Ansan-si, Kyonggi-do
  - Soon Chun Hyang University Bucheon Hospital ( Site 1812), Bucheon-si, Kyonggi-do
  - Hallym University Dongtan Sacred Heart Hospital ( Site 1813), Hwaseong-si, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Internal Medicine ( Site 1803), Suwon, Kyonggi-do
  - Dong-A University Hospital ( Site 1810), Busan, Pusan-Kwangyokshi
  - Kyungpook National University Chilgok Hospital-Division of Infectious Diseases ( Site 1804), Deagu, Taegu-Kwangyokshi
  - Chungnam national university hospital ( Site 1814), Junggu, Taejon-Kwangyokshi
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 1802), Seoul
  - Asan Medical Center ( Site 1809), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 1806), Seoul
  - Hallym University Kangnam Sacred Heart Hospital ( Site 1807), Seoul
  - Ewha Womans University Mokdong Hospital-Infectious Diseases ( Site 1805), Seoul
  - Korea University Guro Hospital ( Site 1800), Seoul
- Spain (6):
  - EBA CENTELLES ( Site 1100), Centelles, Catalonia
  - Hospital Universitario Getafe ( Site 1111), Getafe, Madrid, Comunidad de
  - Fundación Oftalmologica del Mediterraneo-Vaccine Research ( Site 1118), Valencia, Valenciana, Comunitat
  - Centre d'Atenció Primària Vallcarca - Sant Gervasi ( Site 1101), Barcelona
  - EAP Sardenya ( Site 1102), Barcelona
  - Hospital La Princesa-Clinical Pharmacology ( Site 1115), Madrid
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital-Infectious diseases Division, Department of, Kaohsiung City
  - National Cheng Kung University Hospital ( Site 1901), Tainan
  - National Taiwan University Hospital ( Site 1900), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 1902), Taoyuan District
- Turkey (Türkiye) (5):
  - Sancaktepe Şehit Prof.Dr. İlhan Varank Eğitim ve Arastirma Hastanesi ( Site 1305), Sancaktepe, Istanbul
  - ANKARA UNIVERSITY IBNI SINA HOSPITAL ( Site 1304), Ankara
  - Hacettepe Universite Hastaneleri-İnfection ( Site 1300), Ankara
  - Gazi University Health Research and Application Center Gazi Hospital-Enfeksiyon Hastalıkları ( Site, Ankara
  - Acibadem Universitesi Atakent Hastanesi-Infectious Disease ( Site 1301), Istanbul
- United Kingdom (6):
  - Accellacare - Yorkshire-MeDiNova Yorkshire ( Site 1405), Shipley, Bradford
  - Barts Health NHS Trust-William Harvey Clinical Research Centre ( Site 1407), London, England
  - Royal Free Hospital-Ian Charleson Day Centre RESEARCH ( Site 1402), London, England
  - Layton Medical Centre ( Site 1400), Blackpool, Lancashire
  - Accellacare - Northamptonshire ( Site 1403), Corby, Northamptonshire
  - Accellacare - Warwickshire ( Site 1404), Coventry, Warwickshire

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Jotterand V, Jagannath V, Diaz AA, Velez JD, Letica A, Perez SN, Clark R, Caraco Y, Degen O, Park KH, Unal S, Wittke F, Hurtado K, Churchill C, Zhang Y, Fernsler D, Li J, Buchwald UK, Platt H. A Phase 3 Randomized Trial Investigating the Safety, Tolerability, and Immunogenicity of V116, an Adult-Specific Pneumococcal Vaccine, Compared with PPSV23, in Adults >/=50 Years of Age (STRIDE-10). Vaccines (Basel). 2025 Mar 22;13(4):341. doi: 10.3390/vaccines13040341. PMID 40333240
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26201&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1484 participants were randomized in the base study. Additionally, a subgroup of the first 700 participants randomized in the base study to either V116 or PPSV23 were followed for an additional 18 months after completing Visit 5 as part of an immunogenicity substudy extension. 80 participants enrolled at selected study sites were followed for an additional 6 months after completing Visit 5 as part of a PBMC substudy extension. These substudies investigated exploratory objectives.
Groups:
- V116: Participants received a single intramuscular (IM) vaccination of 0.5 mL of V116 on Day 1 in the base study. Selected participants were followed for an additional 18 months as a part of the immunogenicity substudy extension. Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.
- PPSV23: Participants received a single IM vaccination of 0.5 mL of PPSV23 on Day 1 in the Base Study. Selected participants were followed for an additional 18 months as a part of the immunogenicity substudy extension. Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.
Period: Base Study
Arm/Group | V116 | PPSV23
Started (All Randomized Participants) | 741 | 743
Vaccinated (All Participants as Treated (APaT)) | 739 | 741
Completed | 733 | 735
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Immunogenicity Substudy Extension
Arm/Group | V116 | PPSV23
Started | 350 (Selected participants were followed for an additional 18 months as a part of an immunogenicity substudy extension.) | 350 (Selected participants were followed for an additional 18 months as a part of an immunogenicity substudy extension.)
Completed | 335 | 338
Not Completed | 15 | 12
Not completed — Lost to Follow-up | 3 | 4
Not completed — Randomized by mistake without study treatment | 0 | 2
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Non-Study pneumococcal vaccine administered | 0 | 1
Period: PBMC Substudy Extension
Arm/Group | V116 | PPSV23
Started | 41 (Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.) | 39 (Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.)
Completed | 39 | 39
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Base Study: V116: Participants received a single intramuscular (IM) vaccination of 0.5 mL of V116 on Day 1.
- Base Study: PPSV23: Participants received a single IM vaccination of 0.5 mL of PPSV23 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Base Study: V116 | Base Study: PPSV23 | Total
Number analyzed (Participants) | 741 | 743 | 1484
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.4) | 63.7 (8.3) | 63.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 333 | 665
  Male | 409 | 410 | 819
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 151 | 162 | 313
  Not Hispanic or Latino | 579 | 571 | 1150
  Unknown or Not Reported | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 151 | 140 | 291
  Native Hawaiian or Other Pacific Islander | 9 | 3 | 12
  Black or African American | 2 | 2 | 4
  White | 455 | 469 | 924
  More than one race | 119 | 124 | 243
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consisted of pain/tenderness, redness/erythema, and swelling. 95% confidence intervals (CIs) for between-group differences are provided using the Miettinen & Nurminen method.
Time Frame: Up to 5 days postvaccination
Population: All randomized participants that received a vaccination. Participants are included in the group corresponding to the vaccination received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants
  Injection site erythema | 4.7 | 6.3
  Injection site pain | 39.0 | 35.2
  Injection site swelling | 4.9 | 4.3
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Injection site erythema: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = -1.6, 95% CI 2-sided [-4.0 to 0.7] — V116 minus PPSV23
Statistical Analysis 2: Comparison: Base Study: V116 vs Base Study: PPSV23; Injection site pain: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = 3.7, 95% CI 2-sided [-1.2 to 8.7] — V116 minus PPSV23
Statistical Analysis 3: Comparison: Base Study: V116 vs Base Study: PPSV23; Injection site swelling: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = 0.6, 95% CI 2-sided [-1.6 to 2.7] — V116 minus PPSV23

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs consist of the following: fatigue (tiredness), headache, myalgia (muscle aches), and pyrexia (maximum temperature ≥ 100.4 °F/38.0 °C). 95% confidence intervals (CIs) for between-group differences are provided using the Miettinen & Nurminen method.
Time Frame: Up to 5 days postvaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants
  Fatigue | 16.5 | 15.7
  Headache | 13.7 | 12.0
  Myalgia | 5.3 | 5.9
  Pyrexia | 1.1 | 1.3
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Fatigue: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = 0.9, 95% CI 2-sided [-2.9 to 4.6] — V116 minus PPSV23
Statistical Analysis 2: Comparison: Base Study: V116 vs Base Study: PPSV23; Headache: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = 1.7, 95% CI [-1.8 to 5.1] — V116 minus PPSV23
Statistical Analysis 3: Comparison: Base Study: V116 vs Base Study: PPSV23; Myalgia: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = -0.7, 95% CI [-3.1 to 1.7] — V116 minus PPSV23
Statistical Analysis 4: Comparison: Base Study: V116 vs Base Study: PPSV23; Pyrexia: estimated difference in percent; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = -0.3, 95% CI [-1.5 to 0.9] — V116 minus PPSV23

3. Primary Outcome: Percentage of Participants With Vaccine-Related Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an other important medical event. SAEs that were reported to be at least possibly related by the investigator to study vaccination are summarized. 95% confidence intervals (CIs) for between-group differences are provided using the Miettinen & Nurminen method.
Time Frame: Up to 6 months postvaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants | 0 | 0
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Vaccine-Related Serious Adverse Events; Test type: Other — Estimated difference in percent and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Difference in Percent = 0.0, 95% CI [-0.5 to 0.5] — V116 minus PPSV23

4. Primary Outcome: Serotype-Specific Opsonophagocytic (OPA) Geometric Mean Titers (GMTs) for All Serotypes in V116
Description: Serotype-specific OPA titers for all serotypes in V116 following vaccination were determined using multiplex opsonophagocytic assay (MOPA). Serotype-specific OPA GMTs and GMT ratios with 95% confidence intervals (CIs), and they hypothesis test (1-sided p-value), were calculated using a constrained longitudinal data analysis (cLDA) model. Per protocol, within-group CIs, or any other method of dispersion were not planned or calculated.
Time Frame: Day 30 postvaccination
Population: Per protocol, all randomized participants who were vaccinated and were without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint and who had sufficient data to perform the analysis. Deviations include, but are not limited to the following: randomized but not vaccinated, blood drawn out of time window, prohibited concomitant medication or vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Titers
  3: number analyzed (Participants) | 725 | 729
  3 | 230.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 211.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  7F: number analyzed (Participants) | 729 | 732
  7F | 4876.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3314.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  8: number analyzed (Participants) | 730 | 733
  8 | 3379.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2882.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  9N: number analyzed (Participants) | 728 | 729
  9N | 7346.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6545.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  10A: number analyzed (Participants) | 725 | 726
  10A | 4382.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2818.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  11A: number analyzed (Participants) | 728 | 729
  11A | 3711.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1809.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  12F: number analyzed (Participants) | 728 | 732
  12F | 3031.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1854.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  17F: number analyzed (Participants) | 722 | 730
  17F | 8215.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4060.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  19A: number analyzed (Participants) | 731 | 732
  19A | 2670.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1879.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  20A: number analyzed (Participants) | 730 | 733
  20A | 6966.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4208.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  22F: number analyzed (Participants) | 725 | 728
  22F | 4724.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3084.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  33F: number analyzed (Participants) | 727 | 731
  33F | 15497.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 17483.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  6A: number analyzed (Participants) | 729 | 730
  6A | 3193.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 964.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15A: number analyzed (Participants) | 715 | 703
  15A | 6746.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1462.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15C: number analyzed (Participants) | 729 | 730
  15C | 7604.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2605.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  16F: number analyzed (Participants) | 726 | 723
  16F | 6675.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1482.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23A: number analyzed (Participants) | 711 | 690
  23A | 4804.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 837.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23B: number analyzed (Participants) | 730 | 726
  23B | 2252.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 137.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  24F: number analyzed (Participants) | 723 | 705
  24F | 4568.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1346.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  31: number analyzed (Participants) | 730 | 731
  31 | 5040.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 423.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  35B: number analyzed (Participants) | 728 | 732
  35B | 10707.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1735.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 3: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — A conclusion of non-inferiority is based on the lower bound of the 95% CI for the estimated GMT ratio (V116/PPSV23) being >0.5 (one-sided p-value <0.025); p < 0.001, cLDA model — 1-sided; GMT Ratio = 1.09, 95% CI 2-sided [0.96 to 1.23] — V116/PPSV23
Statistical Analysis 2: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 7F: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 1.47, 95% CI 2-sided [1.29 to 1.68] — V116/PPSV23
Statistical Analysis 3: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 8: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 1.17, 95% CI 2-sided [1.04 to 1.32] — V116/PPSV23
Statistical Analysis 4: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 9N: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 1.12, 95% CI [1.00 to 1.26] — V116/PPSV23
Statistical Analysis 5: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 10A: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.55, 95% CI 2-sided [1.37 to 1.77] — V116/PPSV23
Statistical Analysis 6: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 11A: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 2.05, 95% CI [1.82 to 2.31] — V116/PPSV23
Statistical Analysis 7: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 12F: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.63, 95% CI 2-sided [1.40 to 1.90] — V116/PPSV23
Statistical Analysis 8: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 17F: V116/PPSV23GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 2.02, 95% CI 2-sided [1.77 to 2.31] — V116/PPSV23
Statistical Analysis 9: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 19A: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.42, 95% CI 2-sided [1.26 to 1.60] — V116/PPSV23
Statistical Analysis 10: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 20A: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.66, 95% CI 2-sided [1.46 to 1.88] — V116/PPSV23
Statistical Analysis 11: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 22F: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.53, 95% CI 2-sided [1.34 to 1.75] — V116/PPSV23
Statistical Analysis 12: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 33F: V116/PPSV23 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 0.89, 95% CI 2-sided [0.76 to 1.04] — V116/PPSV23
Statistical Analysis 13: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 6A: V116/PPSV23 GMT Ratio; Test type: Superiority — A conclusion of superiority is based on the lower bound of the 95% CI for the estimated GMT ratio (V116/PPSV23) being >2.0 (one-sided p-value <0.025); p < 0.001, cLDA model — 1-sided; GMT Ratio = 3.31, 95% CI 2-sided [2.84 to 3.87] — V116/PPSV23
Statistical Analysis 14: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15A: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 4.61, 95% CI 2-sided [3.99 to 5.33] — V116/PPSV23
Statistical Analysis 15: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15C: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 2.92, 95% CI [2.50 to 3.42] — V116/PPSV23
Statistical Analysis 16: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 16F: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 4.50, 95% CI 2-sided [3.99 to 5.09] — V116/PPSV23
Statistical Analysis 17: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23A: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 5.74, 95% CI 2-sided [4.81 to 6.85] — V116/PPSV23
Statistical Analysis 18: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23B: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 16.42, 95% CI 2-sided [13.46 to 20.03] — V116/PPSV23
Statistical Analysis 19: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 24F: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 3.39, 95% CI [2.97 to 3.87] — V116/PPSV23
Statistical Analysis 20: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 31: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 11.89, 95% CI 2-sided [10.16 to 13.91] — V116/PPSV23
Statistical Analysis 21: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 35B: V116/PPSV23 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 13]; p < 0.001, cLDA model — 1-sided; GMT Ratio = 6.17, 95% CI 2-sided [5.54 to 6.87] — V116/PPSV23

5. Primary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Serotype-Specific OPAs for Serotypes Unique to V116
Description: The percentage of participants with ≥4-fold rise from baseline in serotype-specific OPAs for the unique pneumococcal serotypes contained in V116 was determined. The 9 unique pneumococcal serotypes in V116 are as follows: 6A, 15A, 15C, 16F, 23A, 23B, 24F, 31, and 35B. Per protocol, within-group CIs, or any other method of dispersion were not planned or calculated.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants
  6A | 79.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 53.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15A | 69.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 30.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15C | 87.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 76.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  16F | 63.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 20.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23A | 70.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 34.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23B | 86.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 44.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  24F | 50.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 14.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  31 | 74.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 18.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  35B | 63.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 6A: V116-PPSV23 Percentage Difference; Test type: Superiority — A conclusion of superiority is based on the lower bound of the 95% CI for the difference [V116 - PPSV23] between the percentages of participants with a ≥4-fold rise from baseline to 30 days postvaccination being >10 percentage points (1-sided p-value <0.025); p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 26.0, 95% CI 2-sided [20.9 to 31.0] — V116 minus PPSV23
Statistical Analysis 2: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15A: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 39.4, 95% CI 2-sided [33.6 to 44.8] — V116 minus PPSV23
Statistical Analysis 3: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15C: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.214, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 11.7, 95% CI 2-sided [7.5 to 15.9] — V116 minus PPSV23
Statistical Analysis 4: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 16F: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 42.9, 95% CI 2-sided [37.8 to 47.8] — V116 minus PPSV23
Statistical Analysis 5: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23A: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 35.9, 95% CI [29.6 to 41.8] — V16 minus PPSV23
Statistical Analysis 6: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23B: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 42.4, 95% CI 2-sided [37.6 to 47.0] — V116 minus PPSV23
Statistical Analysis 7: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 24F: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 35.9, 95% CI [30.6 to 41.0] — V116 minus PPSV23
Statistical Analysis 8: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 31: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 56.2, 95% CI 2-sided [51.5 to 60.5] — V116 minus PPSV23
Statistical Analysis 9: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 35B: V116-PPSV23 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen method — 1-sided; Percent Difference = 58.7, 95% CI [54.6 to 62.7] — V116 minus PPSV23

6. Secondary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Serotype-Specific Cross-Reactive OPAs
Description: OPA induced by serotypes 6A and 15C in V116 but cross-reactive to serotypes 6C and 15B, respectively, were measured. The percentage of participants with ≥4-fold rise from baseline in serotype-specific cross-reactive OPAs was determined. Point estimate, 95% CI, and p-value are based on the Clopper-Pearson method. Per protocol, this outcome measure was not planned or analyzed in the PPSV23 study arm.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: Per protocol, all randomized participants who were vaccinated with V116 and were without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint and who had sufficient data to perform the analysis. Deviations include, but are not limited to: randomized but not vaccinated, blood drawn out of time window, prohibited concomitant medication or vaccination. Per protocol, this outcome measure was not planned or analyzed in the PPSV23 study arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 0
Percentage of Participants
  6C: number analyzed (Participants) | 620 | 0
  6C | 52.7 [48.7 to 56.7] |
  15B: number analyzed (Participants) | 588 | 0
  15B | 72.6 [68.8 to 76.2] |
Statistical Analysis 1: Comparison: Base Study: V116; Serotype 6C; Test type: Other — A conclusion of acceptability is based on the lower bound of the 95% CI of the percentages of participants with a ≥4 fold rise from baseline to 30 days postvaccination being >50 percentage points (1-sided p-value <0.025); p = 0.093, Clopper-Pearson method — 1-sided
Statistical Analysis 2: Comparison: Base Study: V116; Serotype 15B; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, Clopper-Pearson method — 1-sided

7. Secondary Outcome: Serotype-Specific Geometric Mean Fold Rise (GMFR) of OPA GMTs for All Serotypes in V116
Description: The GMFR from baseline in serotype-specific OPA GMTs for all serotypes in V116 was determined using MOPA. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Ratio
  3: number analyzed (Participants) | 595 | 586
  3 | 7.5 [6.8 to 8.3] | 6.8 [6.2 to 7.5]
  7F: number analyzed (Participants) | 641 | 648
  7F | 18.3 [15.8 to 21.1] | 14.0 [12.2 to 16.1]
  8: number analyzed (Participants) | 663 | 671
  8 | 34.3 [29.6 to 39.8] | 28.8 [25.1 to 33.0]
  9N: number analyzed (Participants) | 611 | 602
  9N | 11.3 [10.0 to 12.8] | 11.4 [10.1 to 12.8]
  10A: number analyzed (Participants) | 621 | 618
  10A | 16.6 [14.3 to 19.1] | 10.9 [9.5 to 12.4]
  11A: number analyzed (Participants) | 630 | 643
  11A | 18.5 [15.7 to 21.7] | 9.2 [7.9 to 10.8]
  12F: number analyzed (Participants) | 667 | 669
  12F | 89.2 [78.1 to 101.8] | 58.1 [50.5 to 66.8]
  17F: number analyzed (Participants) | 592 | 609
  17F | 25.2 [21.7 to 29.3] | 12.9 [11.3 to 14.8]
  19A: number analyzed (Participants) | 674 | 682
  19A | 10.2 [9.1 to 11.4] | 7.2 [6.5 to 8.0]
  20A: number analyzed (Participants) | 680 | 680
  20A | 10.9 [9.7 to 12.2] | 6.6 [5.9 to 7.3]
  22F: number analyzed (Participants) | 603 | 616
  22F | 20.5 [17.4 to 24.1] | 12.3 [10.5 to 14.3]
  33F: number analyzed (Participants) | 597 | 604
  33F | 8.8 [7.8 to 10.0] | 10.2 [9.0 to 11.6]
  6A: number analyzed (Participants) | 626 | 626
  6A | 19.5 [16.9 to 22.4] | 5.5 [4.8 to 6.3]
  15A: number analyzed (Participants) | 522 | 524
  15A | 10.4 [9.0 to 12.1] | 2.4 [2.1 to 2.7]
  15C: number analyzed (Participants) | 627 | 634
  15C | 49.4 [42.4 to 57.6] | 17.3 [15.1 to 19.8]
  16F: number analyzed (Participants) | 604 | 616
  16F | 7.0 [6.3 to 7.8] | 1.8 [1.6 to 1.9]
  23A: number analyzed (Participants) | 476 | 426
  23A | 13.9 [11.7 to 16.5] | 2.7 [2.2 to 3.2]
  23B: number analyzed (Participants) | 649 | 632
  23B | 53.9 [45.9 to 63.3] | 4.5 [3.9 to 5.2]
  24F: number analyzed (Participants) | 551 | 507
  24F | 5.5 [4.8 to 6.3] | 1.6 [1.4 to 1.8]
  31: number analyzed (Participants) | 655 | 652
  31 | 19.5 [16.7 to 22.8] | 1.7 [1.5 to 1.9]
  35B: number analyzed (Participants) | 660 | 678
  35B | 7.0 [6.3 to 7.8] | 1.1 [1.1 to 1.2]

8. Secondary Outcome: Serotype-Specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for All Serotypes in V116
Description: The GMCs for serotype-specific IgG antibodies for all serotypes in V116 were determined using pneumococcal electrochemiluminescence (PnECL). The GMC ratio estimation and 95% CI were calculated using a cLDA method. Per protocol, within-group CIs, or any other method of dispersion were not planned or calculated.
Time Frame: Day 30 postvaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: μg/mL
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
μg/mL
  3: number analyzed (Participants) | 731 | 734
  3 | 0.79 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.69 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  7F: number analyzed (Participants) | 731 | 734
  7F | 9.35 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.02 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  8: number analyzed (Participants) | 731 | 734
  8 | 13.83 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 11.85 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  9N: number analyzed (Participants) | 731 | 734
  9N | 11.21 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7.23 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  10A: number analyzed (Participants) | 731 | 734
  10A | 15.05 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7.41 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  11A: number analyzed (Participants) | 731 | 734
  11A | 8.83 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4.01 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  12F: number analyzed (Participants) | 731 | 734
  12F | 2.28 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.14 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  17F: number analyzed (Participants) | 731 | 374
  17F | 16.39 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.85 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  19A: number analyzed (Participants) | 731 | 734
  19A | 9.54 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.42 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  20A: number analyzed (Participants) | 731 | 734
  20A | 22.97 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 12.32 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  22F: number analyzed (Participants) | 731 | 734
  22F | 5.32 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3.00 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  33F: number analyzed (Participants) | 731 | 734
  33F | 19.12 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 15.70 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  6A: number analyzed (Participants) | 731 | 734
  6A | 5.79 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.53 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15A: number analyzed (Participants) | 731 | 734
  15A | 17.98 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2.01 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15C: number analyzed (Participants) | 731 | 734
  15C | 19.27 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.61 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  16F: number analyzed (Participants) | 731 | 734
  16F | 3.48 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.35 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23A: number analyzed (Participants) | 731 | 734
  23A | 4.21 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.56 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23B: number analyzed (Participants) | 731 | 734
  23B | 5.74 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.20 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  24F: number analyzed (Participants) | 731 | 734
  24F | 8.52 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.40 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  31: number analyzed (Participants) | 731 | 734
  31 | 3.48 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.40 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
  35B: number analyzed (Participants) | 731 | 734
  35B | 22.26 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.43 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 3: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.14, 95% CI 2-sided [1.04 to 1.25] — V116/PPSV23
Statistical Analysis 2: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 7F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.86, 95% CI 2-sided [1.65 to 2.10] — V116/PPSV23
Statistical Analysis 3: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 8: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.17, 95% CI 2-sided [1.04 to 1.31] — V116/PPSV23
Statistical Analysis 4: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 9N: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.55, 95% CI 2-sided [1.37 to 1.76] — V116/PPSV23
Statistical Analysis 5: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 10A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 2.03, 95% CI 2-sided [1.79 to 2.31] — V116/PPSV23
Statistical Analysis 6: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 11A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 2.20, 95% CI 2-sided [1.97 to 2.46] — V116/PPSV23
Statistical Analysis 7: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 12F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.99, 95% CI 2-sided [1.72 to 2.30] — V116/PPSV23
Statistical Analysis 8: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 17F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 2.39, 95% CI 2-sided [2.12 to 2.70] — V116/PPSV23
Statistical Analysis 9: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 19A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.49, 95% CI 2-sided [1.32 to 1.67]; V116/PPSV23
Statistical Analysis 10: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 20A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.86, 95% CI 2-sided [1.65 to 2.10] — V116/PPSV23
Statistical Analysis 11: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 22F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.77, 95% CI 2-sided [1.55 to 2.02] — V116/PPSV23
Statistical Analysis 12: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 33F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 1.22, 95% CI 2-sided [1.08 to 1.37] — V116/PPSV23
Statistical Analysis 13: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 6A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 3.78, 95% CI 2-sided [3.29 to 4.35] — V116/PPSV23
Statistical Analysis 14: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 8.92, 95% CI 2-sided [7.89 to 10.09] — V116/PPSV23
Statistical Analysis 15: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 15C: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 3.43, 95% CI 2-sided [3.01 to 3.92] — V116/PPSV23
Statistical Analysis 16: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 16F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 9.84, 95% CI 2-sided [8.83 to 10.97] — V116/PPSV23
Statistical Analysis 17: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23A: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 7.59, 95% CI 2-sided [6.68 to 8.61] — V116/PPSV23
Statistical Analysis 18: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 23B: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 4.79, 95% CI 2-sided [4.26 to 5.38] — V116/PPSV23
Statistical Analysis 19: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 24F: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 21.19, 95% CI [18.98 to 23.65] — V116/PPSV23
Statistical Analysis 20: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 31: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 8.69, 95% CI 2-sided [7.82 to 9.65] — V116/PPSV23
Statistical Analysis 21: Comparison: Base Study: V116 vs Base Study: PPSV23; Serotype 35B: V116/PPSV23 GMC Ratio; Test type: Other — GMCs, GMC ratio, and 95% CI are estimated from a cLDA model; GMC Ratio = 15.53, 95% CI 2-sided [14.13 to 17.07] — V116/PPSV23

9. Secondary Outcome: Serotype-Specific GMFR of IgG GMCs for All Serotypes in V116
Description: The GMFR from baseline in GMCs for serotype-specific IgG antibodies for all serotypes in V116 was determined using PnECL. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Ratio
  3: number analyzed (Participants) | 709 | 715
  3 | 5.3 [5.0 to 5.8] | 4.7 [4.4 to 5.0]
  7F: number analyzed (Participants) | 710 | 716
  7F | 19.3 [17.5 to 21.4] | 10.9 [10.0 to 11.8]
  8: number analyzed (Participants) | 710 | 716
  8 | 16.4 [14.9 to 18.1] | 14.1 [13.0 to 15.3]
  9N: number analyzed (Participants) | 710 | 716
  9N | 20.1 [18.1 to 22.4] | 13.3 [12.2 to 14.5]
  10A: number analyzed (Participants) | 710 | 716
  10A | 22.3 [20.2 to 24.7] | 11.1 [10.2 to 12.1]
  11A: number analyzed (Participants) | 710 | 716
  11A | 10.9 [9.8 to 12.0] | 5.0 [4.7 to 5.4]
  12F: number analyzed (Participants) | 710 | 716
  12F | 20.5 [18.4 to 22.9] | 10.6 [9.5 to 11.7]
  17F: number analyzed (Participants) | 710 | 716
  17F | 25.5 [23.1 to 28.1] | 10.8 [9.9 to 11.8]
  19A: number analyzed (Participants) | 710 | 716
  19A | 7.8 [7.1 to 8.6] | 5.3 [4.9 to 5.7]
  20A: number analyzed (Participants) | 710 | 716
  20A | 15.8 [14.4 to 17.3] | 8.6 [7.9 to 9.3]
  22F: number analyzed (Participants) | 710 | 716
  22F | 19.1 [17.3 to 21.2] | 11.0 [10.0 to 12.1]
  33F: number analyzed (Participants) | 710 | 716
  33F | 14.4 [13.1 to 15.8] | 12.0 [11.0 to 13.0]
  6A: number analyzed (Participants) | 710 | 716
  6A | 17.1 [15.3 to 19.0] | 4.6 [4.2 to 5.1]
  15A: number analyzed (Participants) | 710 | 716
  15A | 27.5 [24.9 to 30.4] | 3.1 [2.9 to 3.4]
  15C: number analyzed (Participants) | 710 | 716
  15C | 30.1 [27.1 to 33.4] | 8.8 [8.0 to 9.6]
  16F: number analyzed (Participants) | 710 | 716
  16F | 15.4 [14.1 to 16.9] | 1.6 [1.5 to 1.7]
  23A: number analyzed (Participants) | 710 | 716
  23A | 20.4 [18.4 to 22.6] | 2.8 [2.6 to 3.0]
  23B: number analyzed (Participants) | 710 | 716
  23B | 13.3 [12.0 to 14.7] | 2.9 [2.7 to 3.1]
  24F: number analyzed (Participants) | 709 | 716
  24F | 23.0 [20.8 to 25.6] | 1.1 [1.1 to 1.1]
  31: number analyzed (Participants) | 710 | 716
  31 | 13.0 [11.9 to 14.3] | 1.6 [1.5 to 1.7]
  35B: number analyzed (Participants) | 710 | 716
  35B | 16.8 [15.3 to 18.5] | 1.1 [1.0 to 1.1]

10. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise From Baseline in Serotype-Specific OPA GMTs for All Serotypes in V116
Description: The percentage of participants with ≥4-fold rise from baseline in serotype-specific OPA GMTs for all serotypes in V116 was determined with MOPA. The within-group CIs were calculated based on the Clopper-Pearson method.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants
  3: number analyzed (Participants) | 595 | 586
  3 | 69.2 [65.4 to 72.9] | 66.9 [62.9 to 70.7]
  7F: number analyzed (Participants) | 641 | 648
  7F | 75.2 [71.7 to 78.5] | 69.9 [66.2 to 73.4]
  8: number analyzed (Participants) | 663 | 671
  8 | 83.6 [80.5 to 86.3] | 85.4 [82.5 to 88.0]
  9N: number analyzed (Participants) | 611 | 602
  9N | 72.3 [68.6 to 75.9] | 73.3 [69.5 to 76.8]
  10A: number analyzed (Participants) | 621 | 618
  10A | 74.7 [71.1 to 78.1] | 66.5 [62.6 to 70.2]
  11A: number analyzed (Participants) | 630 | 643
  11A | 72.1 [68.4 to 75.5] | 58.8 [54.9 to 62.6]
  12F: number analyzed (Participants) | 667 | 669
  12F | 93.3 [91.1 to 95.0] | 90.7 [88.3 to 92.8]
  17F: number analyzed (Participants) | 592 | 609
  17F | 84.1 [80.9 to 87.0] | 71.8 [68.0 to 75.3]
  19A: number analyzed (Participants) | 674 | 682
  19A | 70.9 [67.3 to 74.3] | 64.1 [60.3 to 67.7]
  20A: number analyzed (Participants) | 680 | 680
  20A | 71.0 [67.5 to 74.4] | 58.1 [54.3 to 61.8]
  22F: number analyzed (Participants) | 603 | 616
  22F | 76.5 [72.9 to 79.8] | 67.2 [63.3 to 70.9]
  33F: number analyzed (Participants) | 597 | 604
  33F | 66.2 [62.2 to 70.0] | 70.9 [67.1 to 74.5]
  6A: number analyzed (Participants) | 626 | 626
  6A | 79.1 [75.7 to 82.2] | 53.0 [49.0 to 57.0]
  15A: number analyzed (Participants) | 522 | 524
  15A | 69.7 [65.6 to 73.6] | 30.3 [26.4 to 34.5]
  15C: number analyzed (Participants) | 627 | 634
  15C | 87.9 [85.1 to 90.3] | 76.2 [72.7 to 79.4]
  16F: number analyzed (Participants) | 604 | 616
  16F | 63.2 [59.3 to 67.1] | 20.3 [17.2 to 23.7]
  23A: number analyzed (Participants) | 476 | 426
  23A | 70.6 [66.3 to 74.6] | 34.7 [30.2 to 39.5]
  23B: number analyzed (Participants) | 649 | 632
  23B | 86.6 [83.7 to 89.1] | 44.1 [40.2 to 48.1]
  24F: number analyzed (Participants) | 551 | 507
  24F | 50.5 [46.2 to 54.7] | 14.6 [11.6 to 18.0]
  31: number analyzed (Participants) | 655 | 652
  31 | 74.4 [70.8 to 77.7] | 18.3 [15.4 to 21.4]
  35B: number analyzed (Participants) | 660 | 678
  35B | 63.8 [60.0 to 67.5] | 5.2 [3.6 to 7.1]

11. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise From Baseline in Serotype-Specific IgG GMCs for All Serotypes in V116
Description: The percentage of participants with ≥4-fold rise from baseline in serotype-specific IgG GMCs for all serotypes in V116 was determined using PnECL. The within-group CIs were calculated based on the Clopper-Pearson method.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: V116 | Base Study: PPSV23
Number analyzed (Participants) | 739 | 741
Percentage of Participants
  3: number analyzed (Participants) | 709 | 715
  3 | 59.8 [56.1 to 63.4] | 54.7 [51.0 to 58.4]
  7F: number analyzed (Participants) | 710 | 716
  7F | 84.8 [81.9 to 87.4] | 79.7 [76.6 to 82.6]
  8: number analyzed (Participants) | 710 | 716
  8 | 84.4 [81.5 to 87.0] | 86.5 [83.7 to 88.9]
  9N: number analyzed (Participants) | 710 | 716
  9N | 85.5 [82.7 to 88.0] | 83.2 [80.3 to 85.9]
  10A: number analyzed (Participants) | 710 | 716
  10A | 88.9 [86.3 to 91.1] | 81.1 [78.1 to 83.9]
  11A: number analyzed (Participants) | 710 | 716
  11A | 76.8 [73.5 to 79.8] | 56.6 [52.8 to 60.2]
  12F: number analyzed (Participants) | 710 | 716
  12F | 86.5 [83.7 to 88.9] | 73.7 [70.4 to 76.9]
  17F: number analyzed (Participants) | 710 | 716
  17F | 91.0 [88.6 to 93.0] | 79.6 [76.5 to 82.5]
  19A: number analyzed (Participants) | 710 | 716
  19A | 63.9 [60.3 to 67.5] | 58.5 [54.8 to 62.2]
  20A: number analyzed (Participants) | 710 | 716
  20A | 85.5 [82.7 to 88.0] | 73.3 [69.9 to 76.5]
  22F: number analyzed (Participants) | 710 | 716
  22F | 85.4 [82.5 to 87.9] | 77.5 [74.3 to 80.5]
  33F: number analyzed (Participants) | 710 | 716
  33F | 83.0 [80.0 to 85.7] | 83.5 [80.6 to 86.2]
  6A: number analyzed (Participants) | 710 | 716
  6A | 81.4 [78.3 to 84.2] | 47.3 [43.6 to 51.1]
  15A: number analyzed (Participants) | 710 | 716
  15A | 91.3 [88.9 to 93.2] | 34.2 [30.7 to 37.8]
  15C: number analyzed (Participants) | 710 | 716
  15C | 90.7 [88.3 to 92.7] | 72.1 [68.6 to 75.3]
  16F: number analyzed (Participants) | 710 | 716
  16F | 83.8 [80.9 to 86.4] | 11.3 [9.1 to 13.9]
  23A: number analyzed (Participants) | 710 | 716
  23A | 85.9 [83.1 to 88.4] | 29.9 [26.6 to 33.4]
  23B: number analyzed (Participants) | 710 | 716
  23B | 78.9 [75.7 to 81.8] | 33.1 [29.7 to 36.7]
  24F: number analyzed (Participants) | 709 | 716
  24F | 88.2 [85.5 to 90.4] | 1.7 [0.9 to 2.9]
  31: number analyzed (Participants) | 710 | 716
  31 | 82.0 [78.9 to 84.7] | 11.6 [9.3 to 14.2]
  35B: number analyzed (Participants) | 710 | 716
  35B | 85.1 [82.2 to 87.6] | 2.1 [1.2 to 3.4]

ADVERSE EVENTS:
Time Frame: Up to 24 months postvaccination.
Description: Nonserious AEs through Day 30 postvaccination and all SAEs and deaths through 6 months were collected and reported for all randomized participants who received a vaccination. As pre-specified in the protocol, there were no safety outcome measures associated with the substudies. Per protocol, beyond 6 months postvaccination, participants in the substudies were only assessed for vaccine-related SAEs, deaths (any cause), and any AEs related to a protocol-specified blood draw.
Groups:
- Immunogenicity Substudy: V116: Participants received a single intramuscular (IM) vaccination of 0.5 mL of V116 on Day 1 in the base study. Selected participants were followed for an additional 18 months as a part of an immunogenicity substudy extension.
- Immunogenicity Substudy: PPSV23: Participants received a single intramuscular (IM) vaccination of 0.5 mL of PPSV23 on Day 1 in the base study. Selected participants were followed for an additional 18 months as a part of an immunogenicity substudy extension.
- PBMC Sub-study: V116: Participants received a single intramuscular (IM) vaccination of 0.5 mL of V116 on Day 1 in the base study. Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.
- PBMC Sub-study: PPSV23: Participants received a single IM vaccination of 0.5 mL of PPSV23 on Day 1 in the Base Study. Selected participants were followed for an additional 6 months as a part of a PBMC substudy extension.
Arm/Group | Base Study: V116 | Base Study: PPSV23 | Immunogenicity Substudy: V116 | Immunogenicity Substudy: PPSV23 | PBMC Sub-study: V116 | PBMC Sub-study: PPSV23
All-Cause Mortality (participants affected / at risk) | 0/741 | 0/743 | 0/349 | 0/348 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 22/739 | 18/741 | 0/349 | 0/348 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 399/739 | 364/741 | 0/349 | 0/348 | 0/41 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: V116 (N=739) | Base Study: PPSV23 (N=741) | Immunogenicity Substudy: V116 (N=349) | Immunogenicity Substudy: PPSV23 (N=348) | PBMC Sub-study: V116 (N=41) | PBMC Sub-study: PPSV23 (N=39)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: V116 (N=739) | Base Study: PPSV23 (N=741) | Immunogenicity Substudy: V116 (N=349) | Immunogenicity Substudy: PPSV23 (N=348) | PBMC Sub-study: V116 (N=41) | PBMC Sub-study: PPSV23 (N=39)
Fatigue (General disorders) | 122 (127) | 118 (119) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 58 (59) | 47 (47) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 301 (303) | 261 (261) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 48 (48) | 32 (32) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 43 (43) | 46 (47) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 124 (139) | 105 (117) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT05569954/Prot_SAP_000.pdf